CLINICAL TRIAL: NCT07154823
Title: A Longitudinal Multi-Center Molecular Biomarker Discovery Registry for Patients With Hematologic Malignancies
Acronym: Aquarius
Status: Recruiting | Type: Observational
Sponsor: Tempus AI (Industry)
Responsible Party: Sponsor
Other Study IDs: TP-CA-009
Record Dates: First submitted 2025-08-19; First posted 2025-09-04 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Acute Myeloid Leukaemia (AML); Follicular Lymphoma ( FL)
Keywords: Hematologic Malignancy; Acute Myeloid Leukemia; AML; Next Generation Sequencing; NGS; Follicular Lymphoma
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Lymphoma, Follicular; Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Blood will be collected at pre-specified baseline, follow-up and progression/recurrence or primary refractory disease timepoints. Leftover tissue and/or bone marrow aspirate may be collected depending on the indication of the cohort from standard of care procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 001: Newly Diagnosed Acute Myeloid Leukemia (AML): Newly diagnosed patients with a primary or secondary diagnosis of Acute Myeloid Leukemia (AML)
  Interventions: Other: None - Observational Study
- Cohort 002: Folicular Lymphoma: Cohort 002 contains four subgroups of Follicular Lymphoma (FL): A: Newly Diagnosed FL on Active Observation; B: Newly Diagnosed High Risk FL; C: Relapsed / Refractory High Risk POD24 FL; D: Transformed FL
  Interventions: Other: None - Observational Study

INTERVENTIONS:
Other: None - Observational Study — There are no interventions in this observational study.

SUMMARY:
The TEMPUS AQUARIUS Study is a non-interventional, longitudinal observational study focused on hematological malignancies. It will collect rich molecular (multi-omic) and clinical data from patient cohorts through serial blood draws and the acquisition of leftover tissue and/or bone marrow aspirates during their routine therapy and disease monitoring. The primary goal is to understand the association between biomarkers and real-world clinical outcomes in these patient populations.

ELIGIBILITY:
All Cohorts Inclusion Criteria:

1. Willing and able to participate in the research and provide biospecimens
2. Willing and able to provide informed consent

Cohort 001 Inclusion:

1. Have documented diagnosis of AML according to the World Health Organization (WHO) classification
2. Secondary AML is allowed

Cohort 002 Inclusion:

1. Histologically confirmed diagnosis of Follicular Lymphoma (Subgroups A-D)
2. Submission of baseline sample representative of current disease per laboratory manual (Subgroups A-D)
3. 002A (Newly Diagnosed Active Observation): On active observation for 6 more or less, or intended for active observation
4. 002B (Newly Diagnosed, High Risk): Intended for first line treatment
5. 002B (Newly Diagnosed, High Risk): Meets the criteria for high risk by any of the following: Follicular Lymphoma Inernational Prognostic Index (FLIPI) High Risk, Groupe d'Etude des Lymphomes Follicularies (GELF) High Tumor Burden, Lactate Dehydrogenase (LDH) above the upper limit of normal (ULN)
6. 002C (Relapsed / Refractory High Risk POD24 FL): Documented progression of disease within 24 months (POD24) of first line follicular lymphoma treatment, prior to second line treatment
7. 002D (Transformed FL): Pathologically confirmed transformation

All Cohorts Exclusion Criteria:

1. Not willing or able to adhere with the study procedures

Cohort 001:

1. Have received any prior therapy intended for standard of care (SoC) treatment of AML

Cohort 002:

1. 002A: Received prior treatment for follicular lymphoma
2. 002A: Diagnosed with High Risk follicular lymphoma by any of the following definitions: FLIPI High Risk, GELF High Tumor Burden, LDH above ULN
3. 002A: Resected patients with NED
4. 002B: Intended for active observation
5. 002B: Received prior treatment for follicular lymphoma

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study is intended to include multiple hematologic malignancies.
Sampling Method: Non-Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2026-01-27 (Actual); Primary Completion 2034-11 (Estimated); Study Completion 2035-11 (Estimated)

PRIMARY OUTCOMES:
To assess biomarker landscape in the progression as well as baseline biospecimen samples and correlate with with real-world outcomes across multiple hematologic indications. | 5 years
  The goal of this biomarker discovery registry is to assess DNA and RNA expression patterns and potential biomarkers in biospecimens collected at baseline and throughout treatment, with the goal of generating hypotheses about predictive markers for therapy selection, prognostic indicators, and potential mechanisms of resistance to standard-of-care therapies across multiple hematologic indications.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Thompson, MD, PhD, FASCO, Principal Investigator — Tempus AI
Locations (3):
- United States (3):
  - The Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Cancer Care Specialists of Reno, Reno, Nevada
  - Taylor Cancer Research Center, Maumee, Ohio

REFERENCES:
- [Background] Dohner H, Wei AH, Appelbaum FR, Craddock C, DiNardo CD, Dombret H, Ebert BL, Fenaux P, Godley LA, Hasserjian RP, Larson RA, Levine RL, Miyazaki Y, Niederwieser D, Ossenkoppele G, Rollig C, Sierra J, Stein EM, Tallman MS, Tien HF, Wang J, Wierzbowska A, Lowenberg B. Diagnosis and management of AML in adults: 2022 recommendations from an international expert panel on behalf of the ELN. Blood. 2022 Sep 22;140(12):1345-1377. doi: 10.1182/blood.2022016867. PMID 35797463
- [Background] Dohner H, DiNardo CD, Appelbaum FR, Craddock C, Dombret H, Ebert BL, Fenaux P, Godley LA, Hasserjian RP, Larson RA, Levine RL, Miyazaki Y, Niederwieser D, Ossenkoppele G, Rollig C, Sierra J, Stein EM, Tallman MS, Tien HF, Wang J, Wierzbowska A, Wei AH, Lowenberg B. Genetic risk classification for adults with AML receiving less-intensive therapies: the 2024 ELN recommendations. Blood. 2024 Nov 21;144(21):2169-2173. doi: 10.1182/blood.2024025409. PMID 39133932
- [Background] Charalampous C, Goel U, Kapoor P, Binder M, Buadi FK, Cook J, Dingli D, Dispenzieri A, Fonder AL, Gertz MA, Gonsalves W, Hayman SR, Hobbs MA, Hwa YL, Kourelis T, Lacy MQ, Leung N, Lin Y, Warsame R, Kyle RA, Rajkumar SV, Kumar SK. Outcomes of patients with primary refractory multiple myeloma in the era of triplet and quadruplet induction therapy. Blood Adv. 2023 Aug 22;7(16):4371-4380. doi: 10.1182/bloodadvances.2023009681. PMID 37603349
- [Background] Kumar S, Paiva B, Anderson KC, Durie B, Landgren O, Moreau P, Munshi N, Lonial S, Blade J, Mateos MV, Dimopoulos M, Kastritis E, Boccadoro M, Orlowski R, Goldschmidt H, Spencer A, Hou J, Chng WJ, Usmani SZ, Zamagni E, Shimizu K, Jagannath S, Johnsen HE, Terpos E, Reiman A, Kyle RA, Sonneveld P, Richardson PG, McCarthy P, Ludwig H, Chen W, Cavo M, Harousseau JL, Lentzsch S, Hillengass J, Palumbo A, Orfao A, Rajkumar SV, Miguel JS, Avet-Loiseau H. International Myeloma Working Group consensus criteria for response and minimal residual disease assessment in multiple myeloma. Lancet Oncol. 2016 Aug;17(8):e328-e346. doi: 10.1016/S1470-2045(16)30206-6. PMID 27511158
- [Background] Reed SC, Croessmann S, Park BH. CHIP Happens: Clonal Hematopoiesis of Indeterminate Potential and Its Relationship to Solid Tumors. Clin Cancer Res. 2023 Apr 14;29(8):1403-1411. doi: 10.1158/1078-0432.CCR-22-2598. PMID 36454121
- [Background] Salam DSDA, Thit EE, Teoh SH, Tan SY, Peh SC, Cheah SC. C-MYC, BCL2 and BCL6 Translocation in B-cell Non-Hodgkin Lymphoma Cases. J Cancer. 2020 Jan 1;11(1):190-198. doi: 10.7150/jca.36954. eCollection 2020. PMID 31892985
- [Background] Clara JA, Sallman DA, Padron E. Clinical management of myelodysplastic syndrome/myeloproliferative neoplasm overlap syndromes. Cancer Biol Med. 2016 Sep;13(3):360-372. doi: 10.20892/j.issn.2095-3941.2016.0043. PMID 27807503
- [Background] Myers RM, Li Y, Barz Leahy A, Barrett DM, Teachey DT, Callahan C, Fasano CC, Rheingold SR, DiNofia A, Wray L, Aplenc R, Baniewicz D, Liu H, Shaw PA, Pequignot E, Getz KD, Brogdon JL, Fesnak AD, Siegel DL, Davis MM, Bartoszek C, Lacey SF, Hexner EO, Chew A, Wertheim GB, Levine BL, June CH, Grupp SA, Maude SL. Humanized CD19-Targeted Chimeric Antigen Receptor (CAR) T Cells in CAR-Naive and CAR-Exposed Children and Young Adults With Relapsed or Refractory Acute Lymphoblastic Leukemia. J Clin Oncol. 2021 Sep 20;39(27):3044-3055. doi: 10.1200/JCO.20.03458. Epub 2021 Jun 22. PMID 34156874
- [Background] Eichhorst B, Hallek M. Prognostication of chronic lymphocytic leukemia in the era of new agents. Hematology Am Soc Hematol Educ Program. 2016 Dec 2;2016(1):149-155. doi: 10.1182/asheducation-2016.1.149. PMID 27913474
- [Background] Kikushige Y. Pathogenesis of chronic lymphocytic leukemia and the development of novel therapeutic strategies. J Clin Exp Hematop. 2020 Dec 15;60(4):146-158. doi: 10.3960/jslrt.20036. Epub 2020 Nov 4. PMID 33148933
- [Background] Thomas M. Pharma and the benefits of Real World Data. Drug Discovery World (DDW). Published November 4, 2021. Accessed May 5, 2023. https://www.ddw-online.com/trends-analysis-pharma-and-the-benefits-of-real-world-data-13702-202111/
- [Background] Office of the Commissioner. Oncology Real World Evidence Program. U.S. Food and Drug Administration. Accessed May 5, 2023. https://www.fda.gov/about-fda/oncology-center-excellence/oncology-real-world-evidence-program
- [Background] Vellanki PJ, Ghosh S, Pathak A, Fusco MJ, Bloomquist EW, Tang S, Singh H, Philip R, Pazdur R, Beaver JA. Regulatory implications of ctDNA in immuno-oncology for solid tumors. J Immunother Cancer. 2023 Feb;11(2):e005344. doi: 10.1136/jitc-2022-005344. PMID 36796877
- [Background] Abbosh C, Birkbak NJ, Swanton C. Early stage NSCLC - challenges to implementing ctDNA-based screening and MRD detection. Nat Rev Clin Oncol. 2018 Sep;15(9):577-586. doi: 10.1038/s41571-018-0058-3. PMID 29968853
- [Background] Grayson N. Real-world data can help make better drugs and do it faster. STAT. Published May 2, 2018. Accessed May 5, 2023. https://www.statnews.com/2018/05/02/real-world-data-drug-development/